CLINICAL TRIAL: NCT04167241
Title: Early Peri-operative Right Ventricle Dysfunction Following Major Lung Resection
Brief Title: Right Ventricle Function After Major Right Lung Resection
Acronym: RIVER
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Principal Investigator, Enrico Giustiniano, Principal Investigator, Humanitas Clinical and Research Center
Other Study IDs: RIVER Trial
Record Dates: First submitted 2019-11-08; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Right Ventricular Dysfunction; Pneumonectomy; Status
Keywords: Right Ventricle Disfunction; Pneumonectomy; Echocardiography
MeSH Terms: conditions — Ventricular Dysfunction, Right | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients submitted to right pneumonectomy or bi-lobectomy: Consecutive, elective surgical patients submitted to right pneumonectomy or bi-lobectomy
  Interventions: Diagnostic Test: Echocardiography

INTERVENTIONS:
Diagnostic Test: Echocardiography — Before and after right pneumonectomy or bi-lobectomy patients will receive echocardiography

SUMMARY:
Major lung resection is associated with high post-operative morbidity and mortality and significant long-term decreased functional capacity, especially due to cardiorespiratory complications.

RV (Right Ventricle) ejection, pulmonary artery pressure and tone are tightly coupled. The RV is exquisitely sensitive to changes in afterload. When pulmonary vascular reserve is compromised RV ejection may be also compromised, increasing right atrial pressure and limiting maximal cardiac output. Acute increase in RV outflow resistance, as may occur with acute pulmonary embolism will cause acute RV dilatation and, by ventricular interdependence, markedly decreased LV (Left Ventricle) compliance, rapidly spiraling to acute cardiogenic shock and death.

Most of the studies on RV function after lung resection are small and have found different results, and sometimes conflicting findings. As far as the investigators know, there are no data on the incidence of the RV dysfunction after major lung resection (pneumonectomy/bilobectomy) and it's not clear if there is some direct association between the RV dysfunction and post-operative complications. If so, early detection of RV dysfunction after major lung resection could provide the opportunity for interventional therapy with consequent possible improvement of these patients' prognosis.

DETAILED DESCRIPTION:
The aim of this study is to identify the incidence of early RV systolic dysfunction (defined as Tricuspid Annular Plane Systolic Excursion (TAPSE) < 17 cm, S' (TDI) < 10 cm/s) and estimate the RV-PA (Right Ventricle-Pulmonary Artery) coupling as indicated by Guazzi et all. (TAPSE/PAPs ratio, where PAPs is the Systolic Pulmonary Artery Pressure) after major lung resection (bilobectomy and pneumonectomy) using echocardiography, and to assess if these modifications (RV dysfunction and RV-PA coupling) may be associated with post-operative cardiopulmonary complications occurring during the hospitalization period. Investigators also intend to evaluate if these changes are associated with impaired functional capacity at 3 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients undergoing right pneumonectomy
* Adults patients undergoing pulmonary bilobectomy

Exclusion Criteria:

* Left pneumonectomy (it will not permit TTE postoperatively)
* Completion pneumonectomy
* Patients suffering from any myocardial disease
* Preceding Pulmonary Embolism
* Pregnancy
* Potential pregnancy
* Patients enrolled into another trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients submitted to right pneumonectomy or bi-lobectomy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-08 (Estimated); Primary Completion 2020-11-07 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of right ventricle disfunction | Immediately after the awakening from general anesthesia (Day 0)
  Incidence of early RV systolic dysfunction (defined as TAPSE < 17 mm, S' (TDI) < 10 cm/s) and estimate the RV-PA coupling as indicated by Guazzi et al. (TAPSE/PAPs ratio mm/mmHg) after major lung resection (bilobectomy and pneumonectomy) using echocardiography.

SECONDARY OUTCOMES:
Post-operative outcome | Within 3rd post-operative day
  Pulmonary failure may be associated with post-operative pulmonary embolism
Right ventricle failure | Within 3rd post-operative day
  RV dysfunction and RV-PA uncoupling may be associated with post-operative pulmonary hypertension occurring during the hospitalization period.
Post-operative quality of life | 3 months, post-operatively
  DASI questionnaire

IPD SHARING:
Plan to Share IPD: Undecided